CLINICAL TRIAL: NCT06684821
Title: Analgesic Efficacy of Epidural Neuroplasty Using Racz Catheter During Lumbar Fixation in Situ for Lumbosacral Spondylolisthesis: A Randomized Controlled Trial
Brief Title: Epidural Neuroplasty Using Racz Catheter During Lumbar Fixation in Situ for Lumbosacral Spondylolisthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR903/10/24
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Analgesic Efficacy; Epidural; Neuroplasty; Racz Catheter; Lumbar Fixation; Lumbosacral Spondylolisthesis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Racz catheter group (Experimental): Patients will undergo epidural neuroplasty using Racz catheter during lumber fixation.
  Interventions: Procedure: Racz catheter
- Control group (Active Comparator): Patients will undergo classic lumber fixation.
  Interventions: Procedure: Classic lumber fixation

INTERVENTIONS:
Procedure: Racz catheter — Patients will undergo epidural neuroplasty using Racz catheter during lumber fixation.
  Arms: Racz catheter group
Procedure: Classic lumber fixation — Patients will undergo classic lumber fixation.
  Arms: Control group

SUMMARY:
This study aims to evaluate the analgesic efficacy of epidural neuroplasty using a Racz catheter during lumber fixation in situ for lumbosacral spondylolisthesis.

DETAILED DESCRIPTION:
Lumbosacral spondylolisthesis, a common neurosurgical disorder, involves the anterior displacement of a vertebra in relation to the one below it. It often leads to back pain and neurologic symptoms.

Epidural lysis of adhesions is a procedure which treat chronic LBP in patients which didn't respond to medical treatments.The technique of Radiofrequency ablation (RFA) uses high-frequency current to produce tissue coagulation and heat. It involves the use of radio waves, applied through a percutaneous probe to generate heat and create a lesion in a spinal sensory nerve

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* Patients suffering from spondylolisthesis grade 0, 1, 2 complaining of low back pain and/or sciatica.

Exclusion Criteria:

* Uncooperative patients.
* Patients in need of discectomy for lumber disc prolapse.
* Patients with severe canal stenosis and in need of spinal laminectomy.
* Contraindications to perform the proper technique e.g., coagulopathy and skin infection.
* Body mass index (BMI) ≥35 kg/m2.
* History of allergy to contrast medium.
* Previously operated traditional spine surgeries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Degree of Disability | 6 month post-procedure
  Degree of Disability will be assessed using Oswestry Low Back Disability Questionnaire: This questionnaire has been designed to give us information as to how back pain has affected a patient's ability to manage everyday life. It consists of 10 questions for each question, there is a possible 5 points (0 for the first answer, 1 for the second answer, etc). Add up the total for the 10 questions and rate them on the scale (0-4 no disability, 5-14 mild disability, 15-24 moderate disability, 25-34 severe disability, 35-50 complete disability). It will be assisted pre-procedure as a baseline, after 1, 2, 4, 6 month post-procedure

SECONDARY OUTCOMES:
Degree of pain | 6 month post-procedure
  Each patient will be instructed about postoperative pain assessment with the visual analogue scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed pre-procedure as baseline, immediately post-procedure, 1, 2, 4, 6 month post-procedure
Degree of patient satisfaction | 6 month post-procedure
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)
Incidence of complications | 6 month post-procedure
  Incidence of complications that may occur during the technique such as (bending of the tip of the needle, shearing of the catheter, misplacement of the catheter, blocking of the catheter, blood aspiration and bleeding in the epidural space, hypotension, migration of the catheter, paresthesia, headache and infection) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Elhamid ASA, Elsharkawy MS, Shaheen MM, Hamama K, Nada A, Abdelraheem TM. Analgesic Efficacy of Epidural Neuroplasty via Racz Catheter During Lumbar Fixation In Situ for Lumbosacral Spondylolisthesis: A Randomized Controlled Trial. Anesthesiol Res Pract. 2026 Jan 6;2026:1031307. doi: 10.1155/anrp/1031307. eCollection 2026. PMID 41503144